CLINICAL TRIAL: NCT06729775
Title: Disentangling the Role of Culture, Life Stage, and Information Design to Facilitate Equity in Data Report Back
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00004829; R01ES036236 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2024-12-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Education, Health
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- adolescence - graphical (Active Comparator): adolescence (10~19 yrs.) that receives a traditional graphical (figures/charts/tables) representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span
- adolescence - art-infused (Active Comparator): adolescence (10~19 yrs.) that receives an environment art representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span
- adolescence - geospatial (Active Comparator): adolescence (10~19 yrs.) that receives a geospatial representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span
- young adults - graphical (Active Comparator): young adults (18-26 yrs.) that receives a traditional graphical (figures/charts/tables) representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span
- young adults - art-infused (Active Comparator): young adults (18-26 yrs.) that receives an environment art representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span
- young adults - geospatial (Active Comparator): young adults (18-26 yrs.) that receives a a geospatial representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span
- adults - graphical (Active Comparator): adults (27 yrs.+) that receives a traditional graphical (figures/charts/tables) representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span
- adults - art-infused (Active Comparator): adults (27 yrs.+) that receives an environment art representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span
- adults - geospatial (Active Comparator): adults (27 yrs.+) that receives a geospatial representation of environmental health/quality data
  Interventions: Other: Data report back preference by life span

INTERVENTIONS:
Other: Data report back preference by life span — Data report back preference by life span.

SUMMARY:
There remains a need for novel research that facilitates RBRR in a manner that raises data and environmental health literacy (D/EHL) and supports communities striving for environmental health and structural change. Rooted in bioethics and building upon trusted and established long-term partnerships and leveraging existing datasets, the project goal is to create and pilot a national model of report back that is centered in the margins and engages diverse rural and urban EJ communities to ensure that RBRR reaches all populations in a manner tailored to their individual needs, including culture, life stage, language, and design.

DETAILED DESCRIPTION:
The goal of this intervention study is to learn if the data report back design type can modify data and environmental health literacy learning outcomes in adolescence (10~19 yrs.), young adults (18-26 yrs.) (110), and adults (27 yrs.+).

The main questions it aims to answer are:

* How does design type: (1) graphical (control), art-infused (treatment 1) and geospatial (treatment 2) influence data and environmental health literacy learning outcomes related to numeracy and data literacy?
* How does design type: (1) graphical (control), art-infused (treatment 1) and geospatial (treatment 2) influence data and environmental health literacy learning outcomes related to knowledge and awareness related to environmental risks?
* How does design type: (1) graphical (control), art-infused (treatment 1) and geospatial (treatment 2) influence data and environmental health literacy learning outcomes related to skills and self-efficacy for environmental action?
* How does design type: (1) graphical (control), art-infused (treatment 1) and geospatial (treatment 2) influence data and environmental health literacy learning outcomes related to engaging in environmental health activities?
* [primary hypothesis or outcome measure 1]?
* [primary hypothesis or outcome measure 2]?

Researchers will compare outcomes related to life span and design type to see if the design type leads to difference data and environmental health literacy learning outcomes by life stage. During analysis, in addition to life stage, participants will also be analyzed by select sociodemographic variables, e.g., income, education, and race/ethnicity.

Participants will be asked to:

* Complete a pre-survey (baseline)
* Complete a post-survey
* Review their randomly assigned repot back design
* Participate in a focus group and answer questions about the design
* At minimum of six months later, participate in an interview

Summary statistics and qualitative summaries of findings will be generated and used to inform interpretation of inferential statistical tests comparing subgroups. Statistical analyses (i.e., Chi square tests, plus Cramér's V, Multivariate analysis of variance (MANOVA), Kruskal-Wallis, and/or Mann-Whitney U tests) will be conducted to determine any significant differences related to (1) numeracy and data literacy, (2) knowledge and awareness related to environmental risks and (3) skills and self-efficacy for environmental action occur by data report back design type and sociodemographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Participants should live in Pinal county, Arizona, Gila county, Arizona, and Cuyahoga county, Ohio.

Exclusion Criteria:

* Individuals living outside of the partnering counties will not be eligible for participation.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1546 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in the mean literacy and numeracy based on questionnaire responses. | From enrollment to the end of treatment at 78 weeks
  Likert scale where one is equivalent to "Disagree Very Strongly" and six is Agree Very Strongly.
Changes from baseline in the mean knowledge and awareness risks based on questionnaire responses. | From enrollment to the end of treatment at 78 weeks
  Likert scale where one is equivalent to "Disagree Very Strongly" and six is Agree Very Strongly.
Changes from baseline in the mean skills and self-efficacy based on questionnaire responses. | From enrollment to the end of treatment at 78 weeks
  Likert scale where one is equivalent to "Disagree Very Strongly" and six is Agree Very Strongly.
Changes from baseline in the mean environmental health engagement based on questionnaire responses. | From enrollment to the end of treatment at 78 weeks
  Likert scale where one is equivalent to "Disagree Very Strongly" and six is Agree Very Strongly.
Number of participants reporting themes related to literacy and numeracy. | From enrollment to the end of treatment at 78 weeks
  This is a qualitative analysis; words will be coded and analyzed to identify themes and sentiment's that arise in individual interviews and across all interviews and focus groups.
Number of participants reporting themes related to knowledge and awareness risks | From enrollment to the end of treatment at 78 weeks
  This is a qualitative analysis; words will be coded and analyzed to identify themes and sentiment's that arise in individual interviews and across all interviews and focus groups.
Number of participants reporting themes related to skills and self-efficacy | From enrollment to the end of treatment at 78 weeks
  This is a qualitative analysis; words will be coded and analyzed to identify themes and sentiment's that arise in individual interviews and across all interviews and focus groups.
Number of participants reporting themes related to environmental health engagement. | From enrollment to the end of treatment at 78 weeks
  This is a qualitative analysis; words will be coded and analyzed to identify themes and sentiment's that arise in individual interviews and across all interviews and focus groups.

CONTACTS AND LOCATIONS:
Overall Officials: Monica D Ramirez-Andreotta, PhD, Environmental Science, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
All data generated, including that used to produce both positive and negative study findings, will be preserved. We will develop a tiered approach for sharing metadata, data summaries, and datasets. In partnership with community-based team members, we will develop a process for external researchers to request access to community datasets in a manner consistent with the policies of each partnering organization. Based on discussions with partnering organizations, metadata for datasets may be posted to an external data repository, which will enable external researchers to identify datasets and initiate a data sharing request. All data sharing requests will require approval by the research team and partnering. If approved, then credentialed access will be provided by the appropriate database administrator to the Data Portal, a HIPAA compliant system. Congruent with UArizona and NIH data sharing policies, all de-identified public data will be shared in a publicly accessible data repository.
Supporting Information: Study Protocol
Time Frame: This project follows a community-first reporting model. Working with community partners, scientific data will be made accessible as soon as possible, and no later than the time of an associated publication or the end of the performance period of the extramural award that generated the data, whichever occurs first. Data will remain in repositories for the length of time congruent with NIH and University of Arizona data sharing policies. The current minimum prescribed by NIH is three years following study closeout.
Access Criteria: Public data will be shared congruent with any redistribution restrictions. A de-identification process for HIPAA-compliant data will be initiated, with input from project partners. All data access will be controlled and credentialed, and made available by a data repository only after approval by the research team and community organizations. All data will be deidentified before publishing to data repositories or completing data sharing requests. Individual data-sharing requests will be evaluated to ensure human research participants' protection, rights, and confidentiality. The process for sharing de-identified environmental and survey data (numerical and spatial) will be articulated in the consent process (an opt-in approach). Sharing geospatial information with external partners will be discussed with the team and a policy will be developed that is aligned with community partners policies.